CLINICAL TRIAL: NCT05396573
Title: A Randomized, Blinded, Positive Control Phase 1b Trial to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 mRNA Chimera Vaccine (RQ3013) in Healthy Adults Completed a Two-dose Primary Series of Inactivated Vaccine
Brief Title: A Phase 1b Trial to Evaluate the Safety and Immunogenicity of a SARS-CoV-2 mRNA Chimera Vaccine Against COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Walvax Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai RNACure Biopharma Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RQ3013-005
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — RQ3013 COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RQ3013 (Experimental)
  Interventions: Biological: RQ3013
- Comirnaty (Active Comparator)
  Interventions: Biological: Comirnaty

INTERVENTIONS:
Biological: RQ3013 — A single dose of 30 μg/0.15 mL, a single dose of 60 μg/0.3 mL
  Arms: RQ3013
Biological: Comirnaty — A single dose of 30 μg/0.3 mL
  Arms: Comirnaty

SUMMARY:
This is a phase 1b, randomized, double-blind, positive control trial in healthy adults, intended to evaluate the safety and immunogenicity profile of RQ3013 in healthy adults primed with a two-dose inactivated vaccine 6-9 months earlier. The study vaccine is administered IM in the upper arm deltoid as single booster shot on day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants 18-59 years and 60 years and older, and both males and females should be included;
2. Participants who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
3. Participants who have been primed with a two-dose inactivated vaccine 6-9 months earlier, and the intervals between the two inactivated vaccines was between 21 and 42 days.
4. For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of the pregnancy test must be negative. Participants must voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).

Exclusion Criteria:

1. Receipt of any COVID-19 prophylactic medication other than a primary series of inactivated vaccine (e.g., receipt history of any approved or under developing COVID-19 vaccines, or other COVID-19 prophylactic medication, etc.), or non-standard primary series of inactivated vaccine;
2. Abnormal vital signs with clinical significance at screening, with systolic blood pressure ≥140 mmHg (≥150 mmHg for participants aged ≥ 60 years) and/or diastolic blood pressure ≥90 mmHg, or axillary body temperature ≥ 37.3°C, or abnormal results of laboratory screening tests which was clinically significant at screening;
3. Known allergy, or history of anaphylaxis or other serious adverse reactions to the study vaccine or its excipients;
4. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
5. History of COVID-19, or history of close contact with confirmed/suspected COVID-19 patients, or positive results for SARS-CoV-2 nucleic acid tests at screening;
6. Administration of antipyretics or painkillers within 24 hours prior to vaccination;
7. Receipt of any live attenuated vaccine within 28 days prior to vaccination, or subunit and inactivated vaccine within 14 days prior to vaccination;
8. Receipt of blood or blood-related products, including immunoglobulins, within 3 months prior to vaccination; or any planned use during the study period.
9. Participants with the following diseases:

   1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
   2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
   3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
   4. Currently suffering from or previously diagnosed with infectious diseases, positive screening results for hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, human immunodeficiency virus antibody；
   5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
   6. Asplenia, or functional asplenia；
   7. Presence of severe, uncontrollable or hospitalization indicated cardiovascular diseases, diabetes, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors, except for history of well-controlled chronic diseases, such as diabetes, hypertension, etc.;
   8. Participants who cannot tolerate venepuncture, or have a history of needle or blood phobia;
   9. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
10. Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
11. History of a major surgery, per the investigator's judgment, within 12 weeks before vaccination, or not achieving full recovery after surgery, or any planned major surgery during the study;
12. Pregnant or lactating females; males whose partner plans to conceive; males or females who plan to donate sperm or eggs;
13. Participating or planning to participate in other clinical trials during the study period;
14. Presence of any underlying disease or condition which, in the opinion of the investigator, may place the participant at unacceptable risk, make the participant unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Immediate AEs within 30 minutes after booster vaccination, solicited local and systemic AEs for within 7 days and unsolicited AEs within 28 days following booster vaccination | within 28 days following booster vaccination

SECONDARY OUTCOMES:
Live virus GMT, GMFR and seroconversion rate against Beta and Omicron strain in serum measured at pre booster dose and day 7, 14, 28 after booster dose | pre booster dose and day 7, 14, 28 after booster dose
Pseudovirus GMT, GMFR and seroconversion rate against SARS-CoV-2 Beta and Omicron strain in serum measured at pre booster dose and day 7, 14, 28 after booster dose | pre booster dose and day 7, 14, 28 after booster dose
GMT, GMFR and seroconversion rate of S-Protein Specific IgGs in serum measured at pre booster dose and day 7, 14, 28 after booster dose | pre booster dose and day 7, 14, 28 after booster dose
Live virus GMT, GMFR and seroconversion rate against Beta and Omicron strain in serum measured at 3, 6, 12 months after booster dose | 3, 6, 12 months after booster dose
Pseudovirus GMT, GMFR and seroconversion rate against SARS-CoV-2 Beta and Omicron strain in serum measured at 3, 6, 12 months after booster dose | 3, 6, 12 months after booster dose
GMT, GMFR and seroconversion rate of S-Protein Specific IgGs in serum measured at 3, 6, 12 months after booster dose | 3, 6, 12 months after booster dose
Changes of safety laboratory measures at day 4 following booster vaccination in comparison to pre-boosting levels | day 4 following booster vaccination
SAEs and AESIs throughout the study | 12 months after vaccination

OTHER OUTCOMES:
Spike protein specific CD4+, CD8+, CD4+IFN-γ+, CD4+IL-2+, CD4+TNFα+, CD4+IL-4+, CD4+IL-13+, CD8+IFN-γ+, CD8+IL-2+, CD8+TNFα+ cytokine profiling (flow cytometry) by flow cytometry at baseline and day 7, 14 after booster | baseline and day 7, 14 after booster
Spike protein specific cytokine responses by enzyme-linked immunospot (ELISPOT) assay, IFN-γ, IL-2, IL-4 at baseline and day 7, 14 after booster | baseline and day 7, 14 after booster
Spike protein specific T memory cell responses: CD4+ and CD8+ TCM(CCR7+CD45RA-), TEM(CCR7-CD45RA-) and TSCM(CCR7+CD45RA+CD95+) at baseline and 28 days, 3, 6 months after booster | baseline and 28 days, 3, 6 months after booster

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yuan, Study Director — Walvax Biotechnology Co., Ltd.